CLINICAL TRIAL: NCT04545151
Title: A Randomised, Double-blind, Placebo Controlled, Parallel Group, Multi-centre Trial in Adult Subjects With Newly Diagnosed Type 1 Diabetes Mellitus Investigating the Effect of Verapamil SR on Preservation of Beta-cell Function (Ver-A-T1D)
Brief Title: Verapamil SR in Adults With Type 1 Diabetes
Acronym: Ver-A-T1D
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ver-A-T1D; 2020-000435-45 (EudraCT Number)
Record Dates: First submitted 2020-08-21; First posted 2020-09-10 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: INNODIA; Typ-1 Diabetes; Verapamil; Beta cell; C-peptide
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Verapamil

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Trial participants and research teams will be blinded to the treatment group for the duration of the trial. The double blinding will be achieved by providing verapamil SR identical placebo tablets.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verapamil SR (Experimental): Eligible participants will be randomised into the Verapamil SR arm and receive instructions on frequency of administration (daily intake). 80 participants on the experimental arm are expected to complete the trial.
  Interventions: Drug: Verapamil SR 120 mg
- Placebo (Placebo Comparator): Eligible participants will be randomised into the placebo arm and receive instructions on frequency of administration (daily intake).
  40 participants on the control arm are expected to complete the trial.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Verapamil SR 120 mg — For use as a test product in this blinded study, the IMP will be modified by re-packaging. The film-coated tablets will be squeezed from their blisters and filled into HDPE Twist-Off bottles. Each bottle will be labeled as required per country requirement. Labels will be blinded.
  Drug administration:
  * from Day 0 to Week 4: 120 mg once daily
  * from Week 4 to Week 8: 240 mg once daily
  * from Week 8 to Month 12: 360 mg once daily
  Other Names: VeraHEXAL KHK 120 mg; Isoptin retard 120 mg
  Arms: Verapamil SR
Drug: Placebo — The matching placebo will be filled into HDPE Twist-Off bottles, in the same way as the verum. Each bottle will be labeled as required per country requirement. Labels will be blinded.
  Drug administration:
  * from Day 0 to Week 4: 120 mg once daily
  * from Week 4 to Week 8: 240 mg once daily
  * from Week 8 to Month 12: 360 mg once daily
  Other Names: Matching Placebo for Verapamil SR 120 mg
  Arms: Placebo

SUMMARY:
This study has been set up within the framework of the INNODIA network. INNODIA is a global partnership between 31 academic institutions, 6 industrial partners, a small sized enterprise and 2 patient organizations, bringing their knowledge and experience together with one common goal: "To fight type 1 diabetes". (www.innodia.eu) The overall aim of INNODIA is to advance in a decisive way how to predict, stage, evaluate and prevent the onset and progression of type 1 diabetes (T1D).

For this, INNODIA has established a comprehensive and interdisciplinary network of clinical and basic scientists, who are leading experts in the field of T1D research in Europe and UK (United Kingdom), with complementary expertise from the areas of immunology, Beta-cell biology, biomarker research and T1D therapy, joining forces in a coordinated fashion with industry partners and two foundations, as well as with all major stakeholders in the process, including regulatory bodies and patients with T1D and their families.

DETAILED DESCRIPTION:
The study is a multicenter, randomized, double-blind, placebo-controlled study in volunteers with newly diagnosed diabetes mellitus type 1 (within 6 weeks after diagnosis).

The purpose of the clinical trial is to confirm the effect of 360mg Verapamil sustained release (SR) administered orally once daily (titrated over the first 3 months from 120 mg to 360 mg) on the preservation of beta-cell function measured as stimulated C-peptide after 12 months compared to placebo.

The study has a cross-over design and a duration of approximately 24 months, consisting of 3 telephone visits and 7 visits at the trial site. The duration of the treatment phase with verapamil is 12 months, and an additional (optional) follow-up visit will be carried out 12 months after completion of the study. The study procedures are identical in all 20 clinical centres across Europe and the UK.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Age ≥18 and <45 at consent
* Must have a diagnosis of T1D of within 6 weeks duration at screening (date of the first insulin injection)
* Must have at least one or more diabetes-related autoantibodies present at screening: GADA, IA-2A and/or ZnT8A
* Must have fasting C-peptide levels ≥100 pmol/L measured at screening
* Be willing to comply with intensive diabetes management

Exclusion Criteria:

* Be immunodeficient or have clinically significant chronic lymphopenia: Leukopenia (< 3,000 leukocytes /µL), neutropenia (<1,500 neutrophils/µL), lymphopenia (<800 lymphocytes/µL), or thrombocytopenia (<100,000 platelets/µL)
* Have active signs or symptoms of acute infection at the time of screening
* Be currently pregnant or lactating, or anticipate getting pregnant during the 12 months study period
* Require use of immunosuppressive agents including chronic use of systemic steroids
* Have evidence of current or past human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C infection
* Have any complicating medical issues or abnormal clinical laboratory results that may interfere with study conduct, or cause increased risk to include pre-existing cardiac disease, chronic obstructive pulmonary disease (COPD), sickle cell disease, neurological, or blood count abnormalities as judged by the investigator
* Have a history of malignancies other than skin
* History of liver insufficiency or laboratory evidence of liver dysfunction with aspartate aminotransferase (AST) or alanine transaminase (ALT) greater than 3 times the upper limits of normal
* History of renal insufficiency or evidence of renal dysfunction with creatinine greater than 1.5 times the upper limit of normal
* Current or ongoing use of non-insulin pharmaceuticals that affect glycaemic control within prior 7 days of screening
* Use of any other investigational drug in the previous 30 days and/or intent on using any investigational drug for the duration of the trial
* Current use of Verapamil or other calcium channel blockers
* Known hypersensitivity to Verapamil or to any of its excipients
* Concomitant medication known for significantly inducing or inhibiting CYP3A4 and/or glycoprotein-P metabolism
* Intake of grapefruit juice, licorice, St.John's Wort, cannabidiol, ginkgo biloba
* Substrate intake of CYP3A4 and/or glycoprotein-P metabolism, as judged by the investigator
* Hypotension (of less than 100mmHg systolic), sick sinus syndrome (except patients with a functioning artificial pacemaker), uncompensated heart failure or severe left ventricular dysfunction; marked bradycardia (less than 50 beats/minute), atrial flutter or atrial fibrillation in the presence of an accessory bypass tract (e.g. Wolff-Parkinson-White syndrome), hypertrophic cardiomyopathy, acute myocardial infarction, attenuated neuromuscular transmission (e.g. by myasthenia gravis, Lambert-Eaton syndrome, advanced Duchenne muscular dystrophy)
* ECG second or third degree atrioventricular block; Incomplete branch block
* Any condition that in the investigator's opinion may adversely affect study participation or may compromise the study results
* Current use of ß-blockers

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Area under the stimulated C-peptide response curve | At 12 months
  The primary objective is to determine the changes in stimulated C-peptide response during the first two hours of a mixed meal tolerance test (MMTT) at baseline and after 12 months for 360mg Verapamil SR administered orally once daily versus placebo.

SECONDARY OUTCOMES:
Area under the stimulated C-peptide response curve | At 3, 6, 9 and 24 months
  The area under the stimulated C-peptide response curve over the first two hours of a mixed meal tolerance test (MMTT)
Proinsulin, Insulin, Pro-IAPP and Proglucagon secretion | At baseline and 3, 6, 9 and 12 months
  Proinsulin, Insulin, Pro-IAPP and Proglucagon secretion during the first two hours of a mixed meal tolerance test (MMTT)
Fasting C-peptide | At 12 months
  To determine the effects of 360mg Verapamil SR administered orally once daily on fasting C-peptide and Dried Blood Spot (DBS) C-peptide measurements over time.
DBS C-peptide | At baseline, week 4, week 8, and 3, 6, and 9 months
  The DBS (Dried blood spot) C-peptide measurements at all observation times
Change in HbA1c | Baseline, 12 and 24 months
  To determine the effects of 360mg Verapamil SR administered orally once daily on HbA1c daily total insulin dose and continous glucose monitoring (CGM) time in range.
Severe hypoglycaemic episodes | Baseline to 12 months
  Number of treatment emergent severe hypoglycaemic episodes. Severe hypoglycaemia denotes severe cognitive impairment requiring external assistance for recovery according to the American Diabetes Association (ADA)
DKA | Baseline to 12 months
  Number of treatment emergent episodes of diabetic ketoacidosis
Change in insulin requirements | Baseline, 12 and 24 months
  Change in insulin requirements, baseline to 12 months as the daily total dose (three days average) in units per kg body weight (BW)
Change in T1D associated autoantibodies | Baseline to 12 months
  Change in T1D associated autoantibodies (GADA, IAA, IA-2A and ZnT8A) from baseline to 12 months
Continous glucose monitoring (CGM) | At Baseline and every 2 weeks prior to each visit (week 4, week 8, and 3, 6, and 9 months)
  Continous glucose monitoring (CGM) time in range (70-140 mg/dL, 3.9-7.8 mmol/L) and (70-180 mg/dL, 3.9-10.0 mmol/L), time above range (>180 mg/dL, >10.0 mmol/L), time below range (<70 mg/dL, < 3.9 mmol/L)

OTHER OUTCOMES:
Quality of life: DTSQs questionnaire | At week 4 , month 6 and month 12.
  Patients' quality of life will be assessed by participant-reported outcome measures (PROMS):
  the Diabetes Treatment Satisfaction Questionnaire - DTSQs
Quality of life: DTSQc questionnaire | At month 12
  Patients' quality of life will be assessed by participant-reported outcome measures (PROMS):
  the Diabetes Treatment Satisfaction Questionnaire - DTSQc
Quality of life: ADDQoL questionnaire | At month 6 and at month 12
  Patients' quality of life will be assessed by participant-reported outcome measures (PROMS):
  · the Audit of Diabetes Dependent Quality of Life - ADDQoL
Quality of life: HypoFear questionnaire | At week 4 , at month 6 and at month 12
  Patients' quality of life will be assessed by participant-reported outcome measures (PROMS): the Hypoglycaemia Fear Survey - HFS

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Pieber, MD, Prof, Principal Investigator — Medical University of Graz; Dayan Colin, MD, Prof, Principal Investigator — Cardiff University
Locations (22):
- Medical University of Graz, Department of Internal Medicine Division of Endocrinology and Metabolism, Graz, Styria, Austria
- Belgium (4):
  - Universitair Ziekenhuis Brussel, Brussels
  - Université Libre de Bruxelles/ Hôpital Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Katholieke Universiteit Leuven, Leuven
- Institut National de la Santé et de la Recherche Médicale, Paris, France
- Germany (2):
  - HKA Hannover, Hanover
  - Universität Ulm, Ulm
- Italy (2):
  - Università Vita-Salute San Raffaele, Milan
  - Università degli Studi di Siena, Siena
- United Kingdom (12):
  - Queen Elizabeth Hospital, Birmingham
  - Southmead Hospital, Bristol
  - Addenbrokes Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - NHS Greater Glasgow and Clyde-Queen Elizabeth University Hospital, Department of Diabetes, Glasgow
  - Bart's Hospital QMUL, London
  - Guy's Hospital, London
  - Queens Medical Centre, Nottingham
  - John Radcliffe Hospital, Oxford
  - OCDEM, John Radcliffe Hospital, Oxford
  - Royal Hallamshire Hospital, Sheffield
  - Singleton Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning after publication of the primary results papers reporting the prespecified endpoints described in the Statistical analysis plan. (no end date)
Access Criteria: Researchers who provide a methodologically sound proposal - and if needed an ethics approval for the project will be able to access the IPD and supporting information. Access will be provided for research projects to achieve aims in the approved proposal at the level of individual data including for meta-analyses.
  Proposals should be directed to the Chief-Investigator (who may consult with other members of the trial team).To gain access, data requestors will need to sign a data access agreement. Data will be made available directly to the person requesting the data.

REFERENCES:
- [Background] Atkinson MA, Eisenbarth GS, Michels AW. Type 1 diabetes. Lancet. 2014 Jan 4;383(9911):69-82. doi: 10.1016/S0140-6736(13)60591-7. Epub 2013 Jul 26. PMID 23890997
- [Background] DiMeglio LA, Evans-Molina C, Oram RA. Type 1 diabetes. Lancet. 2018 Jun 16;391(10138):2449-2462. doi: 10.1016/S0140-6736(18)31320-5. PMID 29916386
- [Background] Lachin JM, McGee P, Palmer JP; DCCT/EDIC Research Group. Impact of C-peptide preservation on metabolic and clinical outcomes in the Diabetes Control and Complications Trial. Diabetes. 2014 Feb;63(2):739-48. doi: 10.2337/db13-0881. Epub 2013 Oct 2. PMID 24089509
- [Background] Sorensen JS, Johannesen J, Pociot F, Kristensen K, Thomsen J, Hertel NT, Kjaersgaard P, Brorsson C, Birkebaek NH; Danish Society for Diabetes in Childhood and Adolescence. Residual beta-Cell function 3-6 years after onset of type 1 diabetes reduces risk of severe hypoglycemia in children and adolescents. Diabetes Care. 2013 Nov;36(11):3454-9. doi: 10.2337/dc13-0418. Epub 2013 Aug 29. PMID 23990516
- [Background] Ovalle F, Grimes T, Xu G, Patel AJ, Grayson TB, Thielen LA, Li P, Shalev A. Verapamil and beta cell function in adults with recent-onset type 1 diabetes. Nat Med. 2018 Aug;24(8):1108-1112. doi: 10.1038/s41591-018-0089-4. Epub 2018 Jul 9. PMID 29988125
- [Background] Yin T, Kuo SC, Chang YY, Chen YT, Wang KK. Verapamil Use Is Associated With Reduction of Newly Diagnosed Diabetes Mellitus. J Clin Endocrinol Metab. 2017 Jul 1;102(7):2604-2610. doi: 10.1210/jc.2016-3778. PMID 28368479
- [Background] Cooper-Dehoff R, Cohen JD, Bakris GL, Messerli FH, Erdine S, Hewkin AC, Kupfer S, Pepine CJ; INVEST Investigators. Predictors of development of diabetes mellitus in patients with coronary artery disease taking antihypertensive medications (findings from the INternational VErapamil SR-Trandolapril STudy [INVEST]). Am J Cardiol. 2006 Oct 1;98(7):890-4. doi: 10.1016/j.amjcard.2006.04.030. Epub 2006 Aug 7. PMID 16996868
- [Background] Chen J, Saxena G, Mungrue IN, Lusis AJ, Shalev A. Thioredoxin-interacting protein: a critical link between glucose toxicity and beta-cell apoptosis. Diabetes. 2008 Apr;57(4):938-44. doi: 10.2337/db07-0715. Epub 2008 Jan 2. PMID 18171713
- [Background] Xu G, Chen J, Jing G, Shalev A. Preventing beta-cell loss and diabetes with calcium channel blockers. Diabetes. 2012 Apr;61(4):848-56. doi: 10.2337/db11-0955. PMID 22442301
- [Background] Seaquist ER, Anderson J, Childs B, Cryer P, Dagogo-Jack S, Fish L, Heller SR, Rodriguez H, Rosenzweig J, Vigersky R. Hypoglycemia and diabetes: a report of a workgroup of the American Diabetes Association and the Endocrine Society. Diabetes Care. 2013 May;36(5):1384-95. doi: 10.2337/dc12-2480. Epub 2013 Apr 15. PMID 23589542
- [Background] Workgroup on Hypoglycemia, American Diabetes Association. Defining and reporting hypoglycemia in diabetes: a report from the American Diabetes Association Workgroup on Hypoglycemia. Diabetes Care. 2005 May;28(5):1245-9. doi: 10.2337/diacare.28.5.1245. No abstract available. PMID 15855602
- [Derived] Wych J, Brunner M, Stenson R, Chmura PJ, Danne T, Mander AP, Mathieu C, Dayan C, Pieber TR. Investigating the effect of verapamil on preservation of beta-cell function in adults with newly diagnosed type 1 diabetes mellitus (Ver-A-T1D): protocol for a randomised, double-blind, placebo-controlled, parallel-group, multicentre trial. BMJ Open. 2024 Nov 28;14(11):e091597. doi: 10.1136/bmjopen-2024-091597. PMID 39613428